CLINICAL TRIAL: NCT01440179
Title: Phase II Two Stage Finding Run-in Study of SAR3419, An Anti-CD19 Antibody-Maytansine Conjugate, Administered as a Single Agent by Intravenous Infusion in Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: SAR3419 in Acute Lymphoblastic Leukemia
Acronym: MYRALL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is stopped due to very modest activity compared to competitors
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFC11603; U1111-1118-0642 (Other: UTN); 2012-002961-36 (EudraCT Number)
Record Dates: First submitted 2011-09-21; First posted 2011-09-26 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Acute Lymphocytic Leukaemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — coltuximab ravtansine

ARMS (1):
- SAR3419 (Experimental): Administered for one to two induction cycles, followed by maintenance cycles up to 6 cycles.
  Interventions: Drug: SAR3419

INTERVENTIONS:
Drug: SAR3419 — Pharmaceutical form: concentrate solution for infusion Route of administration: intravenous

SUMMARY:
Primary Objective:

Participants achieving an Objective Response Rate

Secondary Objectives:

* Response duration
* Progression Free Survival
* Minimal residual disease
* Safety
* Pharmacokinetics

DETAILED DESCRIPTION:
The duration of the study for an individual patient will include:

* The screening period = up to 4 weeks prior to the first administration of SAR3419.
* The treatment period:

  * Induction period = 4 to 8 weeks
  * Maintenance = up to a total maintenance treatment of 6 months
  * A safety follow-up period of 42 days after the last dose.
* Any patient who discontinues the study treatment without disease progression will be followed every 2 months until disease progression, initiation of a new anti-cancer therapy, death or end-of-study date, whatever comes first.

ELIGIBILITY:
Inclusion criteria:

* Previously treated Acute Lymphoblastic Leukemia of B cell origin (including Burkitt's lymphoma) in relapse or primary refractory. Patients in first relapse will be eligible regardless of the first remission duration.
* No more than 3 prior salvage therapies.
* Philadelphia positive patients failing treatment with imatinib mesylate are accepted.
* CD19 positive patients.

Exclusion criteria:

None

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of participants achieving an Objective Response Rate | 4 to 8 weeks

SECONDARY OUTCOMES:
Number of participants with Adverse Events | Up to 1 year
Assessment of PK parameter - maximum concentration (Cmax) | Up to 8 months
Assessment of PK parameter - area under curve (AUC) | Up to 8 months
Assessment of PK parameter - half-life (T1/2) | Up to 8 months
Assessment of PK parameter - clearance | Up to 8 months
Assessment of PK parameter - volume in steady state (Vss) | Up to 8 months
Assessment of minimal residual disease (MRD) | 4 to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- United States (5):
  - Investigational Site Number 840006, Denver, Colorado
  - Investigational Site Number 840003, Nashville, Tennessee
  - Investigational Site Number 840001, Houston, Texas
  - Investigational Site Number 840002, San Antonio, Texas
  - Investigational Site Number 840004, Milwaukee, Wisconsin
- France (6):
  - Investigational Site Number 250006, Amiens
  - Investigational Site Number 250001, Paris
  - Investigational Site Number 250002, Pessac
  - Investigational Site Number 250008, Pierre-Bénite
  - Investigational Site Number 250004, Rennes
  - Investigational Site Number 250005, Strasbourg

REFERENCES:
- [Derived] Carol H, Szymanska B, Evans K, Boehm I, Houghton PJ, Smith MA, Lock RB. The anti-CD19 antibody-drug conjugate SAR3419 prevents hematolymphoid relapse postinduction therapy in preclinical models of pediatric acute lymphoblastic leukemia. Clin Cancer Res. 2013 Apr 1;19(7):1795-805. doi: 10.1158/1078-0432.CCR-12-3613. Epub 2013 Feb 20. PMID 23426279